CLINICAL TRIAL: NCT01481480
Title: A Multicenter, Randomized Controlled Trial Comparing Functional Outcomes After Latissimus Dorsi Tendon Transfer or Partial Arthroscopic Repair of Massive Rotator Cuff Tears
Brief Title: Latissimus Dorsi Tendon Transfer or Partial Arthroscopic Repair of Massive Rotator Cuff Tears
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: University Health Network, Toronto (Other); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16nov2011
Record Dates: First submitted 2011-11-24; First posted 2011-11-29 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Full Thickness Rotator Cuff Tear
Keywords: shoulder; rotator cuff; tendon transfer; arthroscopic repair

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Latissimus dorsi tendon transfer (Experimental): A Latissimus dorsi tendon transfer is performed
  Interventions: Procedure: Latissimus dorsi tendon transfer
- Arthroscopic repair (Active Comparator): An arthroscopic repair is performed
  Interventions: Procedure: Arthroscopic repair

INTERVENTIONS:
Procedure: Latissimus dorsi tendon transfer — Latissimus dorsi tendon transfer
  Arms: Latissimus dorsi tendon transfer
Procedure: Arthroscopic repair — Arthroscopic repair
  Arms: Arthroscopic repair

SUMMARY:
A massive tear of the rotator cuff is a debilitating condition that causes pain, significant impairments in strength, and resultant loss of activity of the affected arm. To our knowledge, there is no Level 1 evidence comparing surgical procedures to treat massive rotator cuff tears. Adding the first randomized controlled trial to will be a substantial contribution to the current body of evidence available in the subject of massive rotator cuff tears. Most studies found in the literature following patients with massive rotator cuff tears are retrospective, have small numbers of patients, offer no control group and do not adequately compare treatment methods.Moreover, there is no consensus from experts regarding which treatment is superior.

Our multicentre orthopaedic study group proposes a multicentre randomized clinical trial prospectively comparing latissimus dorsi tendon transfer to arthroscopic management for the treatment of massive rotator cuff tears. This study will include the use of comprehensive functional, motor and radiographic outcome assessments.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 40 to 65 years of age
* Massive rotator cuff tear, identified by MRI as being greater than 4cm in greatest diameter.
* Provision of informed consent

Exclusion Criteria:

* Absence of functioning latissimus dorsi muscle (assessed by "cough test"
* Absence of subscapularis muscle insertion (assessed by MRI)
* Glenohumeral arthritis of Grade 2 or higher, including evidence of acromio-humeral arthritis
* Acute tears (identifiable injury which precluded symptoms in past 6 months)
* Neurologic injury causing paralysis of affected shoulder girdle/arm
* Limited life expectancy due to significant medical co-morbidity or medical contraindication to surgery (ASA Grade IV or higher)
* Anticipated problems, in the judgement of the investigators, with maintaining follow-up (i.e. patients with no fixed address, patients not mentally competent to give consent, etc.)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-08; Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Constant-Murley score | 2 years
  Constant-Murley score at 2 years

SECONDARY OUTCOMES:
Quick Dash | 2 years
  Quick Dash - limb specific patient outcome measurement

CONTACTS AND LOCATIONS:
Overall Officials: Michael McKee, MD, FRSC(C), Principal Investigator — Unity Health Toronto
Locations (1):
- Toronto Western Hospital, St. Michael's Hospital, Holland Centre, Toronto, Ontario, Canada